CLINICAL TRIAL: NCT02203344
Title: Use of Bispectral Index Monitoring as an Alert to Detect Deep Sedation in Mechanical Ventilated Patients: a Prospective Observational Study
Brief Title: BIS Monitoring to Detect Deep Sedation
Status: Completed | Type: Observational
Sponsor: Capital Medical University (Other)
Collaborators: Beijing Municipal Health Bureau (Other)
Responsible Party: Principal Investigator, Jian-Xin Zhou, Professor, Capital Medical University
Other Study IDs: KY2014-05--013
Record Dates: First submitted 2014-07-28; First posted 2014-07-29 (Estimated); Last update posted 2014-12-30 (Estimated); Status verified 2014-12

CONDITIONS: Disorder; Mental, Sedative; Depressed Level of Consciousness; Mechanical Ventilation Complication; Psychosis Associated With Intensive Care
MeSH Terms: conditions — Consciousness Disorders

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Light sedation: Light sedation is defined as RASS of +1 to -2.
- Deep sedation: Deep sedation is defined as RASS of -3 to -5

SUMMARY:
Studies have shown that prolonged deep sedation is associated with adverse clinical outcomes in adult intensive care unit (ICU) patients. The revised guidelines for management of pain, agitation and delirium by the Society of Critical Care Medicine in 2013 also recommended that adult ICU patients should be maintained at a light level of sedation. The key point in light sedation strategy is the assessment of depth of sedation. At present, sedation is monitored mainly by the subjective clinical score systems, such as the Ramsay Scale, the Riker's Sedation-Agitation Scale (SAS) and the Richmond Agitation-Sedation Scale (RASS). However, the subjective and intermittent nature of these scales instruments has limited their application in light sedation algorithm. Consequently, objective and continuous measurement of the level of sedation would be more desirable in clinical practice. In recent years, objective measures of brain function have been of great interests in the evaluation of sedation level, and bispectral index (BIS) has been the most investigated instrument.

Several studies compared BIS with subjective sedation scales in adult ICU patients, and yielded conflicting results. The different approaches to select BIS value may be the most important reason for these inconsistent agreements between BIS and subjective sedation scales. A formal scheme of subjective assessment of the depth of sedation and level of consciousness should incorporate exerting verbal and physical stimuli and observation of the patient's subsequent responses. Our primary aim is to clarify the diagnostic accuracy of BIS in detecting early deep sedation against the reference standard of subjective scale instrument. We hypothesize that BIS monitoring will provide accurate, subjective and continuous evaluation of deepen sedation.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients are intubated and ventilated within the previous 24 hours, are administered with continuous or intermittent intravenous sedatives and/or analgesics, and are expected to receive mechanical ventilation and sedation for longer than 24 hours

Exclusion Criteria:

* Age under 18 or over 65 years;
* Continuously infusion of muscle relaxants;
* Diagnosed or suspected brain diseases, which including brain trauma, intracranial hemorrhage, stroke, brain tumors, hypoxic-ischemic encephalopathy, epilepsy and meningitis;
* Diagnosed conditions that resulted in a decrease level of consciousness, which including hypoxemia with partial pressure of oxygen in arterial blood less than 60 mmHg, hypotension with systolic blood pressure less than 90 mmHg, hypoglycemia with blood glucose concentration less than 4.1 mmol/L, anemia with hemoglobin concentration less than 70 g/L, and body temperature below 36 °C.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients admitted to a 22-bed general ICU in a University Affiliated Hospital will be screened daily and enrolled consecutively.
Sampling Method: Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2014-08; Primary Completion 2014-11 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
The primary aim of present study is to determine the diagnostic accuracy of BIS monitoring for detecting deep sedation against the reference standard of RASS. | 15 minutes before and after RASS evaluation
  According to RASS evaluation, observations in each time point will be stratified into 2 situations: light sedation (RASS= 0 to -2) and deep sedation (RASS= -3 to -5). Receiver operator characteristic (ROC) curve analysis will be applied to determine the probability of BIS values in predicting deep sedation.

SECONDARY OUTCOMES:
Incidence of deep sedation | 24 hours after establishing of BIS monitoring
Occurrence of deep sedation during day- and night-time | 24 hours after establishing of BIS monitoring
  Day-time is defined as 8AM to 8PM, and night-time as 8PM to 8AM.

CONTACTS AND LOCATIONS:
Overall Officials: Jian-Xin Zhou, MD, Principal Investigator — Capital Medical University
Locations (1):
- Department of Critical Care Medicine, Daxing Teaching Hospital, Capital Medical University, Beijing, Beijing Municipality, China